CLINICAL TRIAL: NCT02590848
Title: Walnuts, Long-Chain Polyunsaturated Fatty Acids and Adolescent Brain Development: A Dietary Intervention
Brief Title: Walnuts, Long-Chain Polyunsaturated Fatty Acids and Adolescent Brain Development
Acronym: WALNUTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CP14/00108
Record Dates: First submitted 2015-10-19; First posted 2015-10-29 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2019-07

CONDITIONS: Vitamin/Nutritional Deficiency; Neurobehavioral Manifestations
Keywords: Walnut intake; Brain development; Nutritional intervention; Healthy adolescents
MeSH Terms: conditions — Malnutrition; Neurobehavioral Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group with no intervention (No Intervention): This group will receive healthy recommendations of eating fresh fruits
- Group with walnut intake (Experimental): This group will receive healthy recommendation of eating fresh fruits + 30 g of walnut kernels per day during 6 months.
  Interventions: Dietary Supplement: Walnut intake

INTERVENTIONS:
Dietary Supplement: Walnut intake — Nutritional intervention: 30g walnut kernels per day
  Arms: Group with walnut intake

SUMMARY:
Background: Adolescence is an important period for brain development as a result of increased synaptic plasticity. Omega-3 polyunsaturated fatty acids (n-3 PUFAs) are essential nutrients for brain development and protection against oxidative stress. Walnuts have the highest n-3 PUFA concentrations of all edible plants.

Objective: The investigators hypothesize that walnut intake will increase n-3 PUFA availability in the body to a level that enhances the development of the brain during adolescence. The technicians will conduct a long-term (6 months) population-based randomized controlled trial in teenagers (n=400 in each arm), and determine the effectiveness of the intervention (30 g of walnut kernels per day, ~1.5g of n-3 PUFA) in enhancing brain development.

Methods: Fieldwork team will contact teenagers and families in collaboration with 20 high schools. Families will receive a basic guide on following a healthy diet in order to ensure implementation and adherence. Brain development outcomes will be measured at baseline and after the intervention. The use of computerized neuropsychological tests will provide the precision required to detect even subtle changes in brain development resulting from the nutritional intervention. Behavioral (socio-emotional) development will be assessed in order to cover a wider picture of brain development. Blood samples will be collected to measure n-3 PUFA levels before and after the intervention in a randomized subsample from both groups (control/ intervention). Linear regression models adjusted for baseline neuropsychological scores will be used to analyze the intervention effect.

Implications: The outcomes of this Project are expected to be a greater understanding of the role of n-3 PUFA intake (walnut) in brain development. A major goal in public health research is to develop cost-effective health recommendations to teenagers.

DETAILED DESCRIPTION:
Adolescence, an important window of opportunity and vulnerability for brain development Although less well studied, adolescence is also a critical period of brain development. The brain undergoes important organizational changes, with the re-emergence of gonadotropin-releasing hormone triggering a cascade of hormone dependent processes. Other biological processes involve epigenetic factors, which are highly sensitive to the environment and may therefore make this period of growth more vulnerable to external insults (Morrison, 2013). Moreover, the prefrontal cortex, which carries out important functions such as internally guided behaviors (control of emotion), logical thinking, working memory and organizing skills (executive function), is the last region of the brain to mature (early-twenties). The synaptic plasticity of the prefrontal cortex is accentuated during adolescence, a process that involves loss of grey matter density, and an increase in white matter volume, cerebral blood flow and synaptic pruning. Adolescence is also a time of refinement of brain connectivity and complex behaviors (Selemon, 2013). It is widely recognized that the synaptic plasticity of the brain decreases with age (Morrison, 2013; Selemon, 2013), but this pattern does not seem to follow a linear trend, and adolescence is an important period during which brain development can be enhanced and protected from environmental hazards with long-term consequences (everything from air pollution to social stress). There is a need for greater understanding of the biological pathways through which the environment affects human brain development, particularly during adolescence, when the most complex behaviors are refined to adulthood sophistication.

Long-chain polyunsaturated fatty acids, walnuts and brain development Nutrition during pregnancy, lactation, childhood and adolescence has a fundamental influence on overall development. Essential fatty acids are long chain polyunsaturated acids (LCPUFAs) that the body cannot synthesize by itself, and must be obtained through the diet (mainly from oily fish, seeds and nuts). Three of these fatty acids play an essential role in brain development: omega-3 (docosahexaenoic (DHA) and eicosapentaenoic (EPA) acids) and omega-6 (arachidonic acid (AA)) (McCann, 2005). LCPUFAs comprise approximately 15 to 30% of the brain's dry weight (Hallahan, 2005), and are involved in the function and architecture of the central nervous system throughout various stages of life. Studies show that DHA regulates neurotransmission systems such as serotonergic, dopaminergic, norepinephrinergic, and acetylcholinergic systems (Fontani, 2005). Of all edible plants, walnuts have the highest level of the omega-3 fatty acid, alpha-linolenic acid (ALA). ALA is the precursor for DHA and EPA, the two most essential fatty acids for the brain (Carey, 2013). Walnuts are also rich in fiber, vitamins, minerals, and other bioactive substances, such as phenolic antioxidants and phytosterols (Bao, 2013). Several studies have confirmed an increment in blood n-3 PUFA levels and improvements in lipid profile after a short-term intervention of a few walnuts per day (Marangoni, 2007; Maranhao, 2011). While most human studies have shown the cardiovascular benefits of walnut intake (Poulose, 2014), there is a need to investigate the potential beneficial effects on brain development, some incipient research on adults show positive results in cognition, these results are further described in Background section (Pribis, 2012; Sánchez-Villegas, 2011). These findings in adults provide a proof of concept for the potential brain development benefits of walnuts, which never has been studied among young teenagers.

This question could be investigated by using a population-based randomized controlled trial to assess whether walnut intake shows beneficial effects on teenage brain function (using neuropsychological assessments). It is ethical and feasible to recommend and facilitate walnut intake (30 g/day; Marangoni, 2007; Maranhao, 2011) over a long period of time (e.g. 12 months; de Ruyter, 2012). A Californian walnut contains ~0.40g of n-3 PUFAs (USDA National Nutrient Database for Standard Reference, 2012), such that a few walnuts (kernel 30g) per day would meet recommendations to consume at least 1g of n-3 PUFAs per day (Food and Nutritional Board, Institute of Medicine of the National Academies, US, 2014). Young Spanish adults (16-25 years) eat about 10g of nuts per day on average (Salas, 2013). Sea food also contains high n-3 PUFA concentrations, but sea food interventions are contra-indicated due to their methylmercury content, an important neurotoxic environmental pollutant (Grandjean, 2014). A limitation of using walnuts is that intake is less consistent than with a daily pill supplement of 1g of DHA, although this specific food recommendation is socially cost-effective and would be complied with by a wider range of people in the global health context.

Neuropsychological and behavioral assessment, using repeated measurements Recent experience in incorporating neuropsychological assessment into our cohort studies from INMA (Environment and Childhood, Guxens, 2012) has resulted in fruitful exchanges of knowledge between neuropsychologists and epidemiologists. Computerized neuropsychological tests performed in repeated exams are the most sensitive tool for studying high-order brain function and development in the general population (Julvez, 2010). Moreover, these tests have been shown in population-based studies to be very sensitive to the effects of environmental and nutritional determinants (Julvez, 2013). The investigators will build on this experience to efficiently select the appropriate range of tests to cover the complex neurofunctions that rapidly develop during adolescence, such as computer tests of working memory, executive function, motor speed, visual reasoning, selective and sustained attention and inhibitory functions (Selemon, 2012). Furthermore, the neuropsychological tests will be complemented by behavioral rating scales aimed at covering the socio-emotional endpoints that are so important during early adolescence (Selemon, 2012; Morrison, 2013). The fact to evaluate other behavioral areas (i.e., social competence and ADHD symptoms) may enrich the interpretation of the findings, and, possibly it contributes to further understand the intrinsic mechanisms. One limitation is the risk of losing outcome consistency because of selecting much dispersed behavioral areas without taking into account the link between them. The best option is a careful selection of neuropsychological and behavioral tools that efficiently embrace several areas of teenage brain development. Only a few trials of n-3 PUFA among adolescents over 11 years have used computer-based neuropsychological tests (Janssen, 2014). A recent large randomized controlled trial among healthy young adults using computerized cognitive tests found that reaction time latencies and working memory were improved after 6 months of DHA supplementation (Stonehouse, 2013). A double-blind, placebo-controlled trial among children with ADHD (7-12 years) found no treatment associations, but in the observational data, a positive association between DHA levels and computerized test scores of divided attention (Milte, 2012) was reported. Large trials measuring neuropsychological functioning using repeated computerized tests within the same subjects have not yet been carried out among healthy young adolescents, and this is required to better understand 'normal' brain development.

The specific hypotheses are:

1. Walnut intake intervention for six months will enhance neuropsychological development among teenagers from general population. The investigators expect to find differences between the two groups (control/walnut) after the intervention.
2. Walnut intake intervention for six months will enhance behavioral (socio-emotional) development among teenagers from general population. The investigators expect to find differences between the two groups after the intervention.
3. Walnut intake intervention for six months will increase n-3 PUFA availability in the body that will be measured in a blood subsample of 200 teenagers at least. The investigators expect to find differences between the two groups (100/100) after the intervention.
4. n-3 PUFA levels in blood will be associated with brain development.

Global Objective The global objective of this population-based randomized controlled trial is to investigate whether the intake of 30 g of walnut kernels (or ~1.5g of n-3 PUFA) per day is beneficial for brain development among teenagers. The combination of sophisticated tools for assessing brain functions, such as computerized neuropsychological tests, will provide the precise data required to detect even subtle changes in brain development resulting from the effects of the nutritional intervention. Further assessments using behavioural rating scales will give us a wider look of the potential effects of the intervention.

Specific objectives

1. Determine the effectiveness of long-term intervention (30g of walnut kernels per day for 6 months) in enhancing neuropsychological development. This project will provide a new understanding of the role of walnut intake (as a surrogate of n-3 PUFA intake) in the brain development of teenagers. This has an important impact for global health interventions due to the affordability of such interventions in diverse societal groups. A major goal in public health research is to develop effective, cost-effective and feasible health recommendations.
2. Determine the effectiveness of long-term intervention (30g of walnut kernels per day for 6 months) in enhancing behavioural development. In combination with neuropsychological (or cognitive) development, teenage behavioural (socio-emotional) development is essential for a wider assessment of brain development.
3. Investigate the effect of the intervention to n-3 PUFA levels in blood and investigate the association between n-3 PUFA levels and brain development. The importance here relies on understanding the potential biological pathway between the intervention and brain development.

Secondary Objectives To assess the association of diet measured by FFQ and adolescent neuropsychological function.

To assess the association of lifestyle habits assessed by general health questionnaire and adolescent neuropsychological function.

To assess the association of ambient air pollution estimated by LUR models and adolescent neuropsychological function.

To assess the association between different behavioral areas during adolescence.

To assess the association between the walnut intervention and biomarkers related to pathways of oxidative stress and inflammatory system and brain function. These biomarkers are related to candidate circulating miRNAs from brain and a panel of metabolites from 5 different classes (acylcarnitines, amino acids, hexoses, phospho-, and sphingolipids and biogenic amines).

METHODOLOGY WALNUTB scientific approach consists of an ambitious randomized controlled trial in a large population-based sample. Sample: The trial will include 400 healthy teenagers in each arm (12-15 year old) from Barcelona city (1,900,000 inhabitants), the participants will be randomly assigned to two groups (intervention & control) and followed up for 6 months (de Ruyter, 2012) with two identical series (before and after the intervention) of multimodal assessments of brain function, and biomarkers of n-3 PUFA. Power calculation for neuropsychological outcomes: Assigning 400 participants each to the intervention and control groups, and six primary outcomes were considered, with a correlation between them of 0.25. The outcomes were considered to have mean 100 and standard deviation 15, as many neuropsychological scores in the general population. The intervention effect to be detected was 3 points. We considered a type-I error of 0.05 and corrected calculations for multiplicity using Benjamini-Hochberg method. A 10% loss of follow-up was assumed. Additionally, we assumed the final models had an R2 of 20%. With all these considerations, the resulting study would have 95% power to detect the association with at least one outcome, 90% to detect at least two, 80% to detect at least 3, 70% to detect at least 4, 55% to detect at least 5 and 31% to detect the association with all six outcomes.

WP 1: The walnut intervention: Design and setting: This trial cannot be blinded due to the nature of the intervention. The control group will receive no intervention, apart from general healthy eating recommendations (as in the intervention group) and follow-up assessments. Recruitment: Nurses will recruit teenagers (n=400 in each arm) in collaboration with 20 high schools from Barcelona. Implementation and Adherence: The investigators will perform age- and gender-stratified random sampling to assign subjects to one of the two groups. All families will receive a basic guide on following a healthy diet in order to ensure implementation and adherence. Families in the intervention group will receive additional instructions on how to encourage the adolescent to eat 30 g of walnuts per day during 6 months, which the investigators will supply for free. The nurses will contact the families every 3 months for a short checking-interview and to administer a food frequency questionnaire (FFQ).

WP 2: Fieldwork and neuropsychological assessment: The investigators will validate and standardize computerized tests to reduce inter-observer variability during assessment and ensure that data are recorded automatically without errors. Moreover, self-reported and internationally validated psychometrical scales will be used to further assess adolescent socio-emotional behaviour. In this project, the investigators will exploit the interaction between neuropsychologists and epidemiologists to test a range of neuropsychological functions that cover the various complex behaviours that are under development during adolescence.

WP 3: Study the intervention effects and the role of omega-3 polyunsaturated fatty acids: In order to investigate the effects of the intervention, valid measures of the outcomes are necessary (WP2), as are valid measures of the intermediate factors, in this case plasma n-3 PUFA levels. Blood samples will be collected at baseline and after the intervention, centrifuged, and plasma samples stored at -80°C until analysis. Statistical Analysis: The following statistical analyses will be carried out: 1) Assess the effect of the intervention on the ratio of n-6 PUFA to n-3 PUFA (n6-n3 ratio) using linear regression models adjusted for baseline levels. 2) Assess the effect of the intervention on brain development, using the method described in 1) above; 3) Assess the effect of n6-n3 ratio on brain development at baseline, and of n6-n3 ratio change on brain development change from baseline to follow-up. 4) Assess the proportion of the effect of the intervention on brain development that is mediated by n6-n3 ratio change. This proportion can be calculated by comparing results from models with and without the mediator. Analyses 1), 2) and 3) (i.e. those involving the intervention) will be based on intention-to-treat, i.e. using intervention (no/yes) regardless of compliance, in order to estimate the effects of the policy (i.e. to encourage eating 30 g of walnuts per day), rather than the effect of walnut consumption.

Time Frame: The investigators expect to do the recruitment and design the intervention and perform a pilot during the first 12 months (ongoing since January 2015), and to implement the intervention and perform follow-up during 12-24 months. The baseline and final assessments will be completed after 24 months (if the investigators include 2015), the total duration of fieldwork is two years and a third year will be needed to perform data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participants with good communication skills
* No twins and siblings included

Exclusion Criteria:

* Adolescents eating walnuts everyday
* Adolescents with supplements of omega-3 fatty acids
* Adolescents with allergy to walnuts

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 730 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
N-back task | 12 months
  It is a computerized test that takes approximately 25 minutes to complete. The stimulus appears in the laptop screen one by one. Children are invited to press a button in the keyboard when the stimulus is the same as the previous one in the 1-back level. In 2-back, they are required to press the button when the stimulus in the screen is the same as the one presented 2 trials back. In 3-back, they had to press when the stimulus is the same as the one presented 3 trials back. The outcome is d: d prime (d') = z (hit rate) - z (false alarm rate)
ANT: Attention Network Test | 12 months
  A test to provide a measure of the efficiency of three different functions of attention: Alerting (the ability to produce and maintain optimal vigilance and performance during tasks), Orienting (involves shifting attention to sensory stimuli) and Executive attention (involves detecting and resolving conflict among responses, error detection and response inhibition). - Alerting (median RT for no cue - median RT for double cue)
  * Orienting (median RT for central cue - median RT for spatial cue)
  * Executive attention (in data base: conflict) (median RT for incongruent - median RT for congruent).
PMA-R: Primary Mental Abilities- Revised | 12 months
  This test aims to asses Fluid Intelligence. This test was finally selected instead of using Trail Making Test. This latter test assesses attention function and executive function already measured by ANT and N-Back.
Roulettes Task | 12 months
  The Roulettes Task assesses risky decision making for rewards (money gain) and punishments (money loss) separately. More specifically, this tasks assesses whether the participant adjusts is risky behavior according to the probabilities and importance of the outcome. It assesses "hot" executive functions (cognition influenced by emotion).
SDQ: Strengths and Difficulties Questionnaire | 12 months
  Twenty-five questions, organized in five separate sub-scales, were used to assess emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and pro-social behavior. Each subscale was scored from 0 to 10. A Total Difficulties Score (TDS) ranging from 0 to 40 was then generated by summing the scores for all scales except the pro-social behavior scale, which is not used to evaluate mental health.
ADHD-DSM-IV form list: Attention Deficit Hyperactivity Disorder DSM-IV form List | 12 months
  The teacher of the child has to do answer 18 questions of multiple choice in order to rate the ADHD of the child. This is a negative scale (higher scores mean more ADHD symptoms). The scores can be transformed in number of symptoms and diagnostic criterion for ADHD and Inattentive and hyperactive subtypes.
Blood concentration of omega-3 and omega-6 fatty acids | 12 months
  Concentrations of docosahexaenoic acid, arachidonic acid, eicosapentaenoic, alpha-linolenic acid will be measured before and after the intervention.
  All measures will be assessed in plasma (The results will be expressed in relative amounts (% of total FAs)).

SECONDARY OUTCOMES:
Height | 12 months
  In centimeters
Weight | 12 months
  In Kilograms
Blood pressure | 12 months
Spirometry | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Julvez Calvo, PhD, Principal Investigator — Fundació Centre de Recerca en Epidemiologia Ambiental, Barcelona, Spain
Locations (1):
- Fundació Centre de Recerca en Epidemiologia Ambiental, Barcelona, Spain

REFERENCES:
- [Derived] Pinar-Marti A, Gignac F, Fernandez-Barres S, Romaguera D, Sala-Vila A, Lazaro I, Ranzani OT, Persavento C, Delgado A, Carol A, Torrent J, Gonzalez J, Roso E, Barrera-Gomez J, Lopez-Vicente M, Boucher O, Nieuwenhuijsen M, Turner MC, Burgaleta M, Canals J, Arija V, Basagana X, Ros E, Salas-Salvado J, Sunyer J, Julvez J. Effect of walnut consumption on neuropsychological development in healthy adolescents: a multi-school randomised controlled trial. EClinicalMedicine. 2023 Apr 6;59:101954. doi: 10.1016/j.eclinm.2023.101954. eCollection 2023 May. PMID 37096186
- [Derived] Julvez J, Gignac F, Fernandez-Barres S, Romaguera D, Sala-Vila A, Ranzani OT, Persavento C, Delgado A, Carol A, Torrent J, Gonzalez J, Roso E, Barrera-Gomez J, Lopez-Vicente M, Garcia-Esteban R, Boucher O, Forns J, Burgaleta M, Sebastian N, Canals J, Arija V, Basagana X, Ros E, Vendrell J, Salas-Salvado J, Sunyer J. Walnuts, Long-Chain Polyunsaturated Fatty Acids, and Adolescent Brain Development: Protocol for the Walnuts Smart Snack Dietary Intervention Trial. Front Pediatr. 2021 Jun 8;9:593847. doi: 10.3389/fped.2021.593847. eCollection 2021. PMID 34169045
- See also: Project Description — https://www.isglobal.org/en/-/estudi-smart-snack
- See also: Project Description — https://smartsnack.isglobal.org/en/home-main-3/